CLINICAL TRIAL: NCT06497972
Title: Assessing the Blood Glucose Response of Novel Wild Rice Enhanced Food Products (ABWE) Study
Brief Title: Blood Glucose Response of Novel Wild Rice Enhanced Food Products (Trial 1)
Acronym: ABWE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dylan MacKay (Other)
Responsible Party: Sponsor-Investigator, Dylan MacKay, Assistant Professor, University of Manitoba
Organization: University of Manitoba (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: HS25756 (B2022:104)
Record Dates: First submitted 2024-07-04; First posted 2024-07-12 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Blood Glucose
Keywords: glycemic response; glycemic control; rice

STUDY DESIGN:
Intervention Model Description: This is Trial 1 of a project that will consist of 2 acute double-blind cross-over trials. The trials will follow the same study design but investigate 2 types of wild rice products. The wild rice products will be provided by the Myera group.
Who Masked: Participant, Investigator
Masking Description: The allocation of this intervention order will be blinded for the investigators and the participants. Treatment will be given blinded names, such as A and B, but it may be possible to determine what each treatment is due to its appearance, however we will not be informing the participants what the treatments are. The study staff who will be preparing and overseeing the treatments may not be blinded due to the different appearances of the treatments. However, the staff that will conduct the trial results analyses will not be un-blinded until the analyses are complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Consumption of the control white bread product (32 grams, 14.4 grams of carbohydrate) (Active Comparator)
  Interventions: Other: White bread (control, 32 grams, 14.4 grams of carbohydrate)
- Consumption of brown rice cake 40 grams (31 grams of carbohydrate) (Experimental)
  Interventions: Other: Brown rice cake
- Consumption of wild rice brown rice blend cake 40 grams (31 grams of carbohydrate) (Experimental)
  Interventions: Other: Wild rice (25%) and brown rice (75%) cake
- Consumption of the control white bread product (66 grams, 31 grams of carbohydrate) (Active Comparator): This arm was conducted after the first three arms in a non-randomized add on session as we identified an issue with the amount of carbohydrate in out comparator being half of what it was supposed to be. This arm provided 66 grams of white bread control product and there will be a minimum of three days separating each visit.
  Interventions: Other: White bread (control, 66 grams, 31 grams of carbohydrate)

INTERVENTIONS:
Other: White bread (control, 32 grams, 14.4 grams of carbohydrate) — 32 grams of white bread, providing 14.4 grams of carbohydrate, which was incorrectly dosed and matched only half the carbohydrate in the rice cakes.
  Arms: Consumption of the control white bread product (32 grams, 14.4 grams of carbohydrate)
Other: Brown rice cake — A 40g rice cake made of 100% brown rice (providing 31 grams of carbohydrate)
  Arms: Consumption of brown rice cake 40 grams (31 grams of carbohydrate)
Other: Wild rice (25%) and brown rice (75%) cake — A 40g rice cake made of a blend of 25% wild rice and 75% brown rice (providing 31 grams of carbohydrate)
  Arms: Consumption of wild rice brown rice blend cake 40 grams (31 grams of carbohydrate)
Other: White bread (control, 66 grams, 31 grams of carbohydrate) — 66 grams of white bread, providing 31 grams of carbohydrate, this arm was added after the mistake in the first control dosing was discovered, so this arm was not randomized and was completed after the first three.
  Arms: Consumption of the control white bread product (66 grams, 31 grams of carbohydrate)

SUMMARY:
The goal of this acute double-blind cross over trial is to test the effects of a wild rice cake product compared to products currently on the market on glycaemic control. The main questions it aims to answer are:

1. What is the effect compared to products currently on the market on glycaemic control?
2. Is the wild rice product palatable?

Participants will:

* consent to attend 4 study visits being 2.5 hours each
* come to each visit fasted for at least 10-12 hours.
* complete a Motivation to Eat VAS following each blood measure

DETAILED DESCRIPTION:
This trial will be an acute double-blind cross-over trial and will investigate 2 types of rice cake products tested against a white bread control. This is the first of the two trials and will be assessing a wild rice cake and a brown rice cake against a control of white bread.

Participants will fast and arrive at the RCFTR between 7:00 and 11:00 am on the session day. They will be provided either of the study treatment based on randomization sequence. Baseline blood glucose (0 min) will be measured twice via finger stick blood sample right before their first bite of the study product, and at 15, 30, 45, 60, 90 and 120 mins after baseline in duplicate. The timer will be started when they take their first bite. VAS will be completed following consumption of the treatments to measure palatability.

The primary objective is to test the effects of a wild rice cake compared to products currently on the market by evaluating factors that influence glycemic response to wild rice in humans, performed via the finger stick blood glucose that will be measured throughout each session as outlined above.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial
* Male or female between 18-50 years old
* BMI range in between 18.9-29.9 kg/m2
* Fasting glucose <5.6 mmol/L
* Usually eat breakfast
* Participant must receive at least two doses of COVID-19 vaccine that have been recognized by Winnipeg Regional Health Authorities.
* In the Investigator's opinion is able and willing to comply with all trial requirements

Exclusion Criteria:

* Fasting glucose ≥ 5.6 mmol/L or <3.5 mmol/L
* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial
* Participants who indicate that they could not finish study treatments within 10 minutes
* Use of medication or supplements that may influence carbohydrate metabolism, including, not limit to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of screening visit
* History of disordered eating, AIDS, hepatitis, a history of clinically important endocrine (including Type I and Type II diabetes mellitus), cardiovascular (including but not limit to atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary or GI disorders
* Intolerance or allergic reaction to rice
* Existing restrictive dietary habits (such a vegan, low carbohydrate/keto) Date and version No: December 12 , 2022, Version 2 Page 7 of 15
* History of hypertension
* History of cancer within the last two years (except for non-melanoma skin cancer)
* Recent history (within 12 month of screening) or current consumption of >14 drinks per week, (1 drink = 12oz of beer, 5oz of wine or 1.5oz distilled spirits)
* Body weight change over 3.5kg for the past 3 months
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks
* Had significant physical trauma or major surgery in the past 3 month or had trauma or major surgery in the past 3 months

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-07-05 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
The effects of different wild rice products compared to products currently on the market on glycaemic control. | Capillary blood glucose will be measured at 0 (baseline) and then 15, 30, 45, 60, 90 and 120 minutes after the first bite of treatment.
  Finger stick blood glucose will be measured throughout each session.

SECONDARY OUTCOMES:
To measure the palatability of the wild rice products following consumption. | VAS measuring palatability will be completed immediately after the consumption of the treatments.
  Visual Analogue Scale (VAS).

CONTACTS AND LOCATIONS:
Overall Officials: Dylan MacKay, PHD, Principal Investigator — University of Manitoba
Locations (1):
- Chronic Disease Innovation Centre, Seven Oaks Hospital, Winnipeg, Manitoba, Canada